CLINICAL TRIAL: NCT01964170
Title: ASP3550 Phase III Study - An Open-Label, Active-Controlled, Parallel-Arm Study, Comparing ASP3550 With Goserelin Acetate in Patients With Prostate Cancer -
Brief Title: A Study to Compare the Effect of ASP3550 With Goserelin in Patients With Prostate Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Astellas Pharma Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 3550-CL-0010
Record Dates: First submitted 2013-10-15; First posted 2013-10-17 (Estimated); Last update posted 2024-10-31 (Actual); Status verified 2024-10

CONDITIONS: Prostate Cancer
Keywords: ASP3550; Prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — acetyl-2-naphthylalanyl-3-chlorophenylalanyl-1-oxohexadecyl-seryl-4-aminophenylalanyl(hydroorotyl)-4-aminophenylalanyl(carbamoyl)-leucyl-ILys-prolyl-alaninamide; Goserelin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- ASP3550 PART 1 and PART 2 (Experimental): Part 1 for 1 year treatment and Part 2 for an extended period of treatment
  Interventions: Drug: degarelix
- Goserelin (Active Comparator): part 1 for 1 year treatment
  Interventions: Drug: Goserelin

INTERVENTIONS:
Drug: degarelix — subcutaneous
  Other Names: ASP3550
  Arms: ASP3550 PART 1 and PART 2
Drug: Goserelin — subcutaneous
  Arms: Goserelin

SUMMARY:
To compare the efficacy and safety of ASP3550 to goserelin acetate in patients with prostate cancer.

DETAILED DESCRIPTION:
This study consists of two parts. The purpose of PART 1 is to test non-inferiority of ASP3550 to goserelin acetate with respect to the cumulative castration rate in terms of serum testosterone when ASP3550 or goserelin acetate is administered for one-year in patients with prostate cancer.

The patients assigned to receive ASP3550 and completed the treatment in PART 1 are eligible for the treatment in PART 2, and will receive ASP3550 maintenance dose subcutaneously for additional term. The long-term safety, efficacy and PK of the continued ASP3550 treatment will be assessed in PART 2.

ELIGIBILITY:
Inclusion Criteria:

* Male patient with histologically confirmed prostate cancer (adenocarcinoma).
* Patient in whom endocrine treatment is indicated. Patient having undergoing prostatectomy or radiotherapy with curative intention and has a rising serum PSA (PSA ≥ 2 ng/mL at screening) may be included.
* Has a serum testosterone level above 2.2 ng/mL at screening.
* Has an Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) score of 0 to 2 at screening.
* Has a serum PSA ≥ 2 ng/mL at screening.
* Has a life expectancy of at least 12 months.

Exclusion Criteria:

* Previous or present endocrine treatment for prostate cancer. Example: surgical castration, GnRH agonists, GnRH antagonists, antiandrogens or oestrogens, and 5α-reductase inhibitors.
* Received a 5α-reductase inhibitor within 25 weeks preceding screening.
* Is a candidate for curative therapy, i.e., radical prostatectomy or radiotherapy within 12 months.
* Has concurrent or a history of poorly controlled severe asthma, anaphylactic reactions, severe urticaria or angioedema.
* Has hypersensitivity towards mannitol.
* Has a marked prolongation of QT/QTc interval (two consecutive increases to >450 ms in QTc interval at retest) at screening.
* Has concurrent or a history of a disease (heart failure, hypokalemia, a family history of QT prolongation syndrome, etc.) that may induce Torsade de Pointes.

Min Age: 20 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 234 (Actual)
Dates: Start 2013-08-13 (Actual); Primary Completion 2015-06-05 (Actual); Study Completion 2016-08-08 (Actual)

PRIMARY OUTCOMES:
Cumulative castration rate of treatment in terms of serum testosterone level | Up to one year of the treatment

SECONDARY OUTCOMES:
Proportion of castrated subjects in terms of serum testosterone level | Up to one year of the treatment
Proportion of castrated subjects in terms of serum testosterone level | Baseline and Days 3, 7, and 28
Changes in serum levels of prostate-specific antigen (PSA) over time | Up to one year of the treatment
Safety assessed by the incidence of adverse events | up to the end of treatment. approximately for 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Principal Investigator — Astellas Pharma Inc
Locations (8):
- Japan (8):
  - Chugoku
  - Chūbu
  - Hokkaido
  - Kansai
  - Kantou
  - Kyushu
  - Shikoku
  - Tōhoku

IPD SHARING:
Plan to Share IPD: Yes
Access to anonymized individual participant level data collected during the study, in addition to study-related supporting documentation, is planned for studies conducted with approved product indications and formulations, as well as products terminated during development. Studies conducted with product indications or formulations that remain active in development are assessed after study completion to determine if Individual Participant Data can be shared. Further details on Astellas' data sharing policy can be found at https://www.clinicaltrials.astellas.com/transparency/.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Access to participant level data is offered to researchers after publication of the primary manuscript (if applicable) and is available as long as Astellas has legal authority to provide the data.
Access Criteria: Researchers must submit a proposal to conduct a scientifically relevant analysis of the study data. The research proposal is reviewed by an Independent Research Panel. If the proposal is approved, access to the study data is provided in a secure data sharing environment after receipt of a signed Data Sharing Agreement.
URL: https://www.clinicaltrials.astellas.com/transparency/

REFERENCES:
- [Derived] Zengerling F, Jakob JJ, Schmidt S, Meerpohl JJ, Blumle A, Schmucker C, Mayer B, Kunath F. Degarelix for treating advanced hormone-sensitive prostate cancer. Cochrane Database Syst Rev. 2021 Aug 5;8(8):CD012548. doi: 10.1002/14651858.CD012548.pub2. PMID 34350976
- [Derived] Ozono S, Tsukamoto T, Naito S, Horie S, Ohashi Y, Uemura H, Yokomizo Y, Fukasawa S, Kusuoka H, Akazawa R, Saito M, Akaza H. Efficacy and safety of 3-month dosing regimen of degarelix in Japanese subjects with prostate cancer: A phase III study. Cancer Sci. 2018 Jun;109(6):1920-1929. doi: 10.1111/cas.13600. Epub 2018 May 23. PMID 29624800
- See also: Link to results on the Astellas Clinical Study Results website — https://astellasclinicalstudyresults.com/study.aspx?ID=310